CLINICAL TRIAL: NCT00650702
Title: A Phase II, Randomized, Masked, Parallel-Group Study of Safety and Preliminary Efficacy of the Punctum Plug Delivery System in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy of Punctum Plug Delivery System in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Acronym: CORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPL GLAU 02
Record Dates: First submitted 2008-03-27; First posted 2008-04-02 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2011-03

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma, ocular hypertension, IOP
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Low Latanoprost-PPDS
  Interventions: Drug: Latanoprost-PPDS
- 2 (Experimental): Medium Latanoprost-PPDS
  Interventions: Drug: Latanoprost-PPDS
- 3 (Experimental): High Latanoprost-PPDS
  Interventions: Drug: Latanoprost-PPDS

INTERVENTIONS:
Drug: Latanoprost-PPDS — Control of IOP compared to baseline for the low dose of Latanoprost-PPDS for 4 months or until loss of efficacy
  Arms: 1
Drug: Latanoprost-PPDS — Control of IOP compared to baseline for the medium dose of Latanoprost-PPDS for 4 months or until loss of efficacy
  Arms: 2
Drug: Latanoprost-PPDS — Control of IOP compared to baseline for the high dose of Latanoprost-PPDS for 4 months or until loss of efficacy
  Arms: 3

SUMMARY:
The purpose of this study is to determine if the Punctum Plug Delivery System (PPDS) is safe and effective in controlling intraocular pressure in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 yrs with open-angle glaucoma or ocular hypertension
* Subjects who have a best-corrected visual acuity of 20/100 or better.

Exclusion Criteria:

* Uncontrolled medical conditions.
* Subjects who wear contact lenses.
* Subjects requiring chronic topical artificial tears, lubricants, and/or requiring any other chronic topical medications.
* Subjects who have a history of chronic or recurrent inflammatory eye disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Artesia, California
  - Sacramento, California
  - Bel Air, Maryland
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Lynbrook, New York
  - High Point, North Carolina
  - Philadelphia, Pennsylvania